CLINICAL TRIAL: NCT05811663
Title: Health Care Use and Costs of Functional Somatic Disorders: A Population-based Study (DanFunD)
Brief Title: Health Care Use and Costs of Functional Somatic Disorders
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: DanFunD direct healthcare
Record Dates: First submitted 2023-03-02; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Bodily Distress Syndrome; Irritable Bowel; Fibromyalgia; Chronic Widespread Pain; Chronic Fatigue Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Fibromyalgia; Chronic Pain; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DanFunD baseline: Data from the DanFunD baseline cohort will be included. It comprises a total of 9,656 (33.7% of the invited participants) men and women aged 18-76 years born in Denmark and living in the Western part of greater Copenhagen.
  Individuals with FSD are identified by means of self-reported questionnaires (n=9,656) and diagnostic research interviews (n=1,590).
  Participants with FSD will be defined as follows:
  FSD operationalised by the Bodily Distress Syndrome single- and multi-organ type will be defined with both self-reported questionnaires and diagnostic interviews.
  Three functional somatic syndromes, i.e. irritable bowel, chronic widespread pain, and chronic fatigue will be defined with questionnaires.
  Severe physical disease will be defined by means of self-report as having received at least one of the following five diagnoses: Cancer, stroke, myocardial infarction, other heart disease, and obstructive pulmonary disease.

SUMMARY:
The goal of this observational case-control study is to learn about direct healthcare use and costs of functional somatic disorders.

The aim of the proposed study is to investigate the use and costs of direct healthcare for individuals with functional somatic disorders.

Researchers will compare direct healthcare use and costs of individuals with functional somatic disorders and compare them with that of healthy controls and individuals with other severe physical disease, respectively.

DETAILED DESCRIPTION:
Functional somatic disorders (FSD) are common conditions characterized by persistent patterns of physical symptoms that cannot be better explained by other physical or mental conditions. The conditions may cause severe impairment for the patients who are often characterized by impaired physical and mental health, lower social status, and poor labour market association.

In 2005, it was estimated that FSD accounted for 3% of hospitalizations and 10-20% of health care expenses in Denmark, and a newer Danish primary care study has shown patients with FSD to have higher annual health care costs compared with conventionally-defined conditions. In foreign nations, studies in clinical samples have shown increased direct and indirect health care costs of FSD which showed a dose-response relationship with severity of the FSD. One Canadian population-based study found increased health care use and costs in children, adolescents, and young adults with a first health record diagnosis of somatic symptom and related disorders. Even though these previous studies provide valuable knowledge to the field of FSD, their methodology may give rise to bias, i.e. inclusion of highly selected patient samples, the use of various diagnostic criteria for defining FSD, and the establishment of FSD by means of self-report. Evidently, studies investigating the socioeconomic burden in terms of direct health care use and costs of FSD in a randomly obtained population-based sample using solid methodology such as validated symptom criteria and diagnostic interviews for establishing FSD are highly lacking.

The objectives of this proposed study are:

To describe and investigate the healthcare use and healthcare costs for individuals with FSD and compare them with

1. individuals without FSD, and
2. individuals with severe physical disease

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* not born in Denmark
* not being a Danish citizen
* pregnancy.

Ages: 18 Years to 76 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data from the DanFunD baseline cohort will be included. For this cohort, a total of 25,368 men and women aged 18-72 years living in the Western part of Greater Copenhagen were randomly obtained from the nationwide Danish registries and invited to participate; 9656 accepted. All of them answered questionnaires about physical symptoms, physical and mental health as well as social components. A stratified sub sample consisting og every tenth participant together with every high score on the symptoms questionnaires were invited to participate in a diagnostic interview performed over telephone by trained family physicians. A total of 2450 were invited and 1590 accepted and participated in the interview.
Sampling Method: Probability Sample
Enrollment: 9656 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Use of primary healthcare resources 10 years before baseline | 10-year period before the day the participant participated in the DanFunD baseline investigation
  Data on use of healthcare in primary care will be extracted from the Danish National Health Service Register for Primary Care. This category will include number of face-to-face consultations in general practise, medical specialists, physiotherapists, chiropractors, and psychologists.
Costs of primary healthcare resources 10 years before baseline | 10-year period before the day the participant participated in the DanFunD baseline investigation
  Data on costs of healthcare in primary care will be extracted from the Danish National Health Service Register for Primary Care. This category will include number of face-to-face consultations in general practise, medical specialists, physiotherapists, chiropractors, and psychologists.
Use of primary healthcare resources 4 years after baseline | 4-year period after the day the participant participated in the DanFunD baseline investigation
  Data on use of healthcare in primary care will be extracted from the Danish National Health Service Register for Primary Care. This category will include number of face-to-face consultations in general practise, medical specialists, physiotherapists, chiropractors, and psychologists.
Costs of primary healthcare resources 4 years after baseline | 4-year period after the day the participant participated in the DanFunD baseline investigation
  Data on costs of healthcare in primary care will be extracted from the Danish National Health Service Register for Primary Care. This category will include number of face-to-face consultations in general practise, medical specialists, physiotherapists, chiropractors, and psychologists.
Use of secondary healthcare resources 10 years before baseline | 10-year period before the day the participant participated in the DanFunD baseline investigation
  Data on use of healthcare in secondary care will be extracted from the National Patient Registry.
Costs of secondary healthcare resources 10 years before baseline | 10-year period before the day the participant participated in the DanFunD baseline investigation
  Data on costs of healthcare in secondary care will be extracted from the National Patient Registry.
Use of secondary healthcare resources 4 years after baseline | 4-year period after the day the participant participated in the DanFunD baseline investigation
  Data on use of healthcare in secondary care will be extracted from the National Patient Registry.
Costs of secondary healthcare resources 4 years after baseline | 4-year period after the day the participant participated in the DanFunD baseline investigation
  Data on costs of healthcare in secondary care will be extracted from the National Patient Registry.
Use of prescription medication 10 years before baseline | 10-year period before the day the participant participated in the DanFunD baseline investigation
  Data on number of prescriptions will be extracted from The Danish Register Prescription Sales.
Costs of prescription medication 10 years before baseline | 10-year period before the day the participant participated in the DanFunD baseline investigation
  Data on costs of prescriptions will be extracted from The Danish Register Prescription Sales.
Use of prescription medication 4 years after baseline | 4-year period after the day the participant participated in the DanFunD baseline investigation
  Data on number of prescriptions will be extracted from The Danish Register Prescription Sales.
Costs of prescription medication 4 years after baseline | 4-year period after the day the participant participated in the DanFunD baseline investigation
  Data on costs of prescriptions will be extracted from The Danish Register Prescription Sales.

CONTACTS AND LOCATIONS:
Overall Officials: Per W Fink, DMSc, Study Chair — Aarhus University Hospital
Locations (1):
- Marie Weinreich Petersen, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petersen MW, Wellnitz KB, Oernboel E, Carstensen TBW, Meinertz Dantoft T, Ahrendt Bjerregaard A, Joergensen T, Fink P. Healthcare use and costs of functional somatic disorder in Denmark: a population-based cohort study (DanFunD). BMJ Public Health. 2025 Dec 17;3(2):e003318. doi: 10.1136/bmjph-2025-003318. eCollection 2025. PMID 41431615